CLINICAL TRIAL: NCT06683768
Title: Safety of Hypertension Medication Therapy in Patient With Naive Hypertension: a Real-world Study in Japan
Brief Title: A Real-world Study of the Safety of Hypertension Medication Therapy in Japanese Patients With Naïve Hypertension
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696AJP03
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: Essential hypertension; High blood pressure
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Monotherapy Cohort: Adult patients with untreated hypertension who initiated antihypertensive monotherapy (excluding angiotensin receptor neprilysin inhibitor [ARNI]).
- Single-pill Combination (SPC) Cohort: Adult patients with untreated hypertension who initiated single-pill combination antihypertensive therapy.

SUMMARY:
This was a non-interventional, secondary use of data, retrospective, cohort study. The data extracted in this study was used as secondary use of collected patient information in the database, Japan Medical Data Survey (JAMDAS), owned by M3 Inc. (Tokyo, Japan). JAMDAS is a database that aggregates medical information and is constructed mainly from electronic medical record information of medical institutions, allowing real-time extraction of information entered in medical records, such as prescription status including drug switching and continuation, laboratory values, clinical evaluation scores, and comorbidities etc.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed with essential hypertension or hypertensive heart/kidney disease at the index date.
2. Sitting systolic blood pressure (sSBP) ≥150 millimeters of mercury (mm Hg) at the index date.
3. At least one prescription of angiotensin-converting enzyme inhibitor (ACEi), angiotensin receptor blocker (ARB), angiotensin receptor neprilysin inhibitor (ARNI), calcium channel blocker (CCB), diuretics, or these SPCs for hypertension at the index date.
4. At least one visit and blood pressure (BP) measurement within 12 weeks from the index date.

Exclusion criteria:

1. Prescription of hypertensive medication including alpha blocker, beta blocker, alpha-beta blocker, aldosterone antagonist, and renin inhibitor within 24 weeks prior to the index date.
2. Initial prescription of two or more antihypertensive medicines either with or without SPCs at the index date.
3. History of hypotension, hyperkalemia, hypokalemia, or hyponatremia, drug-related or otherwise, or renal failure leading to dialysis, stroke, myocardial infarction, heart failure at the index date or within 24 weeks prior to the index date.
4. History of secondary hypertension (renal parenchymal hypertension, renovascular hypertension [unilateral or bilateral renal artery stenosis] coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension, etc.) at any timepoint.
5. Pregnant women at any timepoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 40563 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs) From Initiation of Antihypertensive Treatment to Weeks 8 and 24 Categorized by Type of AE | Week 8 and Week 24
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Weeks 8 and 24 Categorized by Type of AE | Week 8 and Week 24
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Weeks 8 and 24 Categorized by Type of AE | Week 8 and Week 24
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.

SECONDARY OUTCOMES:
Number of Adverse Events (AEs) From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Blood Pressure (BP) Category | Week 24
  BP Categories included Grade I, II, III, and (isolated) systolic hypertension.
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per BP Category | Week 24
  BP Categories included Grade I, II, III, and (isolated) systolic hypertension.
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per BP Category | Week 24
  BP Categories included Grade I, II, III, and (isolated) systolic hypertension. Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Age Group Category | Week 24
  Age group categories:
  * Less than 65 years old
  * 65 to 74 years old
  * 75 years or older
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Age Group Category | Week 24
  Age group categories:
  * Less than 65 years old
  * 65 to 74 years old
  * 75 years or older
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Age Group Category | Week 24
  Age group categories:
  * Less than 65 years old
  * 65 to 74 years old
  * 75 years or older
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Body Mass Index (BMI) Category | Week 24
  BMI categories:
  * BMI <18.5
  * 18.5 ≤ BMI <25
  * 25 ≤ BMI
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per BMI Category | Week 24
  BMI categories:
  * BMI <18.5
  * 18.5 ≤ BMI <25
  * 25 ≤ BMI
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per BMI Category | Week 24
  BMI categories:
  * BMI <18.5
  * 18.5 ≤ BMI <25
  * 25 ≤ BMI
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Estimated Glomerular Filtration Rate (eGFR) Category | Week 24
  eGFR categories:
  * eGFR <30
  * 30 ≤ eGFR <60
  * 60 ≤ eGFR
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per eGFR Category | Week 24
  eGFR categories:
  * eGFR <30
  * 30 ≤ eGFR <60
  * 60 ≤ eGFR
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per eGFR Category | Week 24
  eGFR categories:
  * eGFR <30
  * 30 ≤ eGFR <60
  * 60 ≤ eGFR
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Potassium Level | Week 24
  Potassium (K) levels:
  * K <3.5
  * 3.5 ≤ K <5.5
  * 5.5 ≤ K
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Potassium Level | Week 24
  Potassium (K) levels:
  * K <3.5
  * 3.5 ≤ K <5.5
  * 5.5 ≤ K
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Potassium Level | Week 24
  Potassium (K) levels:
  * K <3.5
  * 3.5 ≤ K <5.5
  * 5.5 ≤ K
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Creatinine Level | Week 24
  Creatinine (Cr) Levels:
  * Cr <1.5
  * 1.5 ≤ Cr
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Creatinine Level | Week 24
  Creatinine (Cr) Levels:
  * Cr <1.5
  * 1.5 ≤ Cr
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Creatinine Level | Week 24
  Creatinine (Cr) Levels:
  * Cr <1.5
  * 1.5 ≤ Cr
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Proteinuria | Week 24
  Proteinuria:
  * Urine protein <30: Negative
  * 30 ≤ Protein urine: Positive
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Proteinuria | Week 24
  Proteinuria:
  * Urine protein <30: Negative
  * 30 ≤ Protein urine: Positive
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE by Proteinuria | Week 24
  Proteinuria:
  * Urine protein <30: Negative
  * 30 ≤ Protein urine: Positive
  Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Number of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Class of Antihypertensive Medication | Week 24
  Antihypertensive medication classes included calcium channel blockers (CCBs), angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), and diuretics.
Number of Patients With AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Class of Antihypertensive Medication | Week 24
  Antihypertensive medication classes included CCBs, ACE inhibitors, ARBs, and diuretics.
Incidence Rate of AEs From Initiation of Antihypertensive Treatment to Week 24 Categorized by Type of AE per Class of Antihypertensive Medication | Week 24
  Antihypertensive medication classes included CCBs, ACE inhibitors, ARBs, and diuretics. Incidence rate was calculated by dividing the number of patients who had an event by the total number of patients.
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 | Weeks 4, 8, and 12
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by BP Category | Weeks 4, 8, and 12
  BP categories included Grade I, II, and III hypertension.
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by Age Group Category | Weeks 4, 8, and 12
  Age group categories:
  * Less than 65 years old
  * 65 to 74 years old
  * 75 years or older
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by BMI Category | Weeks 4, 8, and 12
  BMI categories:
  * BMI <18.5
  * 18.5 ≤ BMI <25
  * 25 ≤ BMI
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by eGFR Category | Weeks 4, 8, and 12
  eGFR categories:
  * eGFR <30
  * 30 ≤ eGFR <60
  * 60 ≤ eGFR
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by Potassium Level | Weeks 4, 8, and 12
  Potassium (K) levels:
  * K <3.5
  * 3.5 ≤ K <5.5
  * 5.5 ≤ K
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by Creatinine Level | Weeks 4, 8, and 12
  Creatinine (Cr) Levels:
  * Cr <1.5
  * 1.5 ≤ Cr
Change in BP From Initiation of Antihypertensive Treatment to Weeks 4, 8, and 12 by Proteinuria | Weeks 4, 8, and 12
  Proteinuria:
  * Urine protein <30: Negative
  * 30 ≤ Protein urine: Positive
Number of Patients who Achieved the BP Goal at Last Visit Categorized by Subgroup | Up to 13 weeks
  The BP goal was 130/80 millimeters of mercury (mm Hg).
  Subgroups:
  * BP Grade
  * Age
  * BMI
  * Estimated glomerular filtration rate (eGFR)
  * Potassium Level
  * Creatinine Level
  * Proteinuria (positive or negative)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States